CLINICAL TRIAL: NCT03426605
Title: A Phase 1 Dose-Escalation Study of LAM-003 in Patients With Acute Myeloid Leukemia
Brief Title: A Study of LAM-003 in Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OrphAI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LAM-003-HEM-CLN02
Record Dates: First submitted 2018-01-05; First posted 2018-02-08 (Actual); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Oncology; Acute Myeloid Leukemia
MeSH Terms: conditions — Neoplasms; Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Open Label, Dose-Escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LAM-003 (Experimental): Open label LAM-003 at three sequentially increasing starting dose levels of 200, 300 and 450 mg.
  Interventions: Drug: Open Label LAM-003

INTERVENTIONS:
Drug: Open Label LAM-003 — LAM-003

SUMMARY:
A Phase 1 Dose-Escalation Study of LAM-003 in Patients with Acute Myeloid Leukemia

DETAILED DESCRIPTION:
This clinical trial is a Phase 1 study evaluating the safety, pharmacokinetics, pharmacodynamics, and antitumor activity of LAM-003 across a range of LAM-003 dose levels when administered to subjects with previously treated relapsed or refractory cute Myeloid Leukemia (AML).

Subjects will self-administer oral LAM-003 either once or twice per day as long as they are safely benefitting from therapy. Cohorts of 3 to 6 subjects will be sequentially enrolled at progressively higher dose levels of LAM-003 using a standard 3+3 dose-escalation design. Based on the pattern of dose-limiting toxicities observed in the first 4 weeks of therapy, escalation will proceed to define a recommended LAM-003 dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women of age ≥18 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
3. Presence of measurable AML that has progressed during or relapsed after prior therapy
4. All acute toxic effects of any prior antitumor therapy resolved to Grade 1.
5. Adequate hepatic profile.
6. Adequate renal function.
7. Adequate coagulation profile.
8. Negative antiviral serology for human immunodeficiency virus (HIV), hepatitis B, and hepatitis C.
9. For female subjects of childbearing potential, a negative serum pregnancy test.
10. For both male and female subjects, willingness to use adequate contraception.
11. Willingness and ability of the subject to comply with study activities.
12. Evidence of a personally signed informed consent document.

Exclusion Criteria:

1. Leukemic blast cell count >50 × 10^9/L before the start of study therapy and despite the use hydroxyurea, cytarabine, and/or cyclophosphamide.
2. Presence of known central nervous system (CNS) leukemia.
3. Presence of another major cancer.
4. Ongoing Grade >1 proliferative or nonproliferative retinopathy.
5. Significant cardiovascular disease or ECG abnormalities.
6. Significant gastrointestinal disease
7. Uncontrolled ongoing infection.
8. Pregnancy or breastfeeding.
9. Major surgery within 4 weeks before the start of study therapy.
10. Subject was a candidate for hematopoietic stem cell transplantation (HSCT).
11. Ongoing severe graft-versus-house disease (GVHD) with Grade ≥2 serum bilirubin, Grade ≥3 skin involvement, or Grade ≥3 diarrhea at the start of study therapy.
12. Prior solid organ transplantation.
13. Ongoing immunosuppressive therapy other than corticosteroids.
14. Use of a strong inhibitor or inducer of cytochrome P450 (CYP) 3A4.
15. Use of a drug known to prolong the cardiac QT interval.
16. Concurrent participation in another therapeutic or imaging clinical trial.
17. Presence of a concomitant medical condition that (in the judgement of the investigator) interferes with the ability of the subject to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Langdon Miller, M.D., Study Director — AI Therapeutics
Locations (6):
- United States (6):
  - Yale University, New Haven, Connecticut
  - University of Maryland, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Hackensack Meridien Health, Hackensack, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Trial information can be found on AI Therapeutics website — http://ai-therapeutics.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted by 6 investigators located in medical centers throughout the United States.
Pre-assignment Details: The study included a screening period (up to 28 days) prior to the study drug administration period. Discontinuation of prior antitumor therapy was required except that subjects with rapidly proliferative disease could receive AML cytoreduction with hydroxyurea, cytarabine, and/or cyclophosphamide before the start of LAM-003 and during Cycle 1 of LAM-003 administration.
Groups:
- LAM-003 200 mg QD: 6 participants were accrued at starting dose level of 200 mg QD.
- LAM-003 300 mg QD: 3 participants were accrued at 300 mg QD.
- LAM-003 450 mg QD: 4 participants were accrued at 450 mg QD. Intrasubject dose escalations were implemented in 1 subject. Subject 006-006 received LAM-003 450 mg QD during Cycles 1 and 2 and received LAM-003 600 mg QD during Cycles 3 and 4.
- LAM-003 600 mg QD: 4 participants were accrued at 600 mg QD. Intrasubject dose escalations were implemented in 2 subjects:
  * Subject 005-011 received LAM-003 600 mg QD during Cycle 1 and received LAM-003 750 mg QD during Cycles 2 and 3.
  * Subject 006-007 received LAM-003 600 mg QD during Cycle 1 and received LAM-003 750 mg QD during Cycle 2.
Period: Overall Study
Arm/Group | LAM-003 200 mg QD | LAM-003 300 mg QD | LAM-003 450 mg QD | LAM-003 600 mg QD
Started | 6 | 3 | 4 | 4
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 3 | 4 | 4
Not completed — AML relapse or progression | 2 | 1 | 2 | 2
Not completed — Treatment failure | 3 | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The study population was generally consistent with the epidemiology of AML.
Groups:
- LAM-003 600 mg QD: 4 Participant were accrued at 600 mg QD. Intrasubject dose escalations were implemented in 2 subjects:
  * Subject 005-011 received LAM-003 600 mg QD during Cycle 1 and received LAM-003 750 mg QD during Cycles 2 and 3.
  * Subject 006-007 received LAM-003 600 mg QD during Cycle 1 and received LAM-003 750 mg QD during Cycle 2.
- Total: Total of all reporting groups
Arm/Group | LAM-003 200 mg QD | LAM-003 300 mg QD | LAM-003 450 mg QD | LAM-003 600 mg QD | Total
Number analyzed (Participants) | 6 | 3 | 4 | 4 | 17
Age, Continuous [Median (Full Range); unit: years] | 71 [39 to 82] | 34 [26 to 65] | 75 [54 to 83] | 67.5 [48 to 73] | 68 [26 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 1 | 6
  Male | 4 | 2 | 2 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 4 | 3 | 4 | 3 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 2 | 4 | 4 | 13
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 3 | 4 | 4 | 17
BMI [Median (Full Range); unit: kg/m^2] | 32.4 [19 to 45] | 27.6 [26 to 29] | 27.5 [24 to 28] | 21.6 [20 to 48] | 27.6 [19 to 48]
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants]
  0 = Fully active | 0 | 0 | 0 | 1 | 1
  1 = Restricted in physically strenuous activity but ambulatory | 5 | 2 | 1 | 2 | 10
  2 = Ambulatory and capable of all self-care but unable to carry out any work activities | 1 | 1 | 3 | 1 | 6
Elevated peripheral blood AML blast % [Median (Full Range); unit: percentage] | 24.75 [2.9 to 89.3] | 41.40 [13.6 to 95.1] | 22.15 [11.9 to 74.0] | 34.05 [4.5 to 97.1] | 30.40 [2.9 to 97.1]
Number of prior anticancer treatment regimens [Median (Full Range); unit: number of treatments] | 3.0 [2 to 6] | 4.0 [2 to 9] | 3.5 [3 to 4] | 4.0 [4 to 5] | 4.0 [2 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: A primary objective was to determine the LAM-003 MTD and/or recommended dosing regimen (RDR) based on the pattern of dose-limiting toxicities (DLTs) in Cycle 1 of therapy. MTD as determined by DLTs.
Time Frame: At the end of the 28-day observation period for Cycle 1.
Population: Participants were considered evaluable for Cycle 1 DLT assessment if they either had a Cycle 1 DLT or completed 21/28 study drug doses during Cycle 1 and were observed ≥4 weeks from the start of study drug administration without having a DLT.
Measure: Number; unit: DLTs
Arm/Group | LAM-003 200 mg QD | LAM-003 300 mg QD | LAM-003 450 mg QD | LAM-003 600 mg QD
Number analyzed (Participants) | 3 | 3 | 3 | 3
DLTs | 0 | 0 | 0 | 0

2. Secondary Outcome: Adverse Event Assessment
Description: Number and percentage of participants with an adverse event (AE).
Time Frame: Weekly during the first 4 weeks and then every 4 weeks for up to 48 weeks.
Population: All participants who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LAM-003 200 mg QD | LAM-003 300 mg QD | LAM-003 450 mg QD | LAM-003 600 mg QD
Number analyzed (Participants) | 6 | 3 | 4 | 4
Participants
  With ≥1 AE | 6 | 3 | 4 | 4
  With ≥1 TEAE | 6 | 3 | 4 | 4
  With ≥1 study-drug-related TEAE | 3 | 2 | 1 | 2
  With ≥1 TEAE of Grade ≥3 | 5 | 3 | 4 | 3
  With ≥1 study-drug-related TEAE of Grade ≥3 | 0 | 0 | 0 | 0
  With ≥1 SAE | 3 | 3 | 3 | 2
  With ≥1 treatment-emergent SAE | 3 | 3 | 3 | 2
  With ≥1 study-drug-related treatment-emergent SAE | 0 | 0 | 0 | 0
  With ≥1 AESI | 0 | 0 | 0 | 0
  With AEs resulting in drug interruption of study drug | 0 | 0 | 1 | 0
  With AEs (other than AML progression) resulting in permanent discontinuation of study drug | 1 | 0 | 0 | 1
  With AEs resulting in death within 30 days from the last dose of study drug | 1 | 1 | 2 | 1

3. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: The pharmacokinetic parameter Cmax was determined in plasma for the active metabolite of LAM-003A and LAM-003 (prodrug)
Time Frame: Cycle 1 Days 1, 2 and 8 (1 cycle = 28 days)
Population: The Pharmacokinetic (PK) population included all evaluable participants who were dosed and had sufficient concentration-time data to estimate at least one of the planned PK parameters, as determined by the study pharmacokineticist.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LAM-003 200 mg QD | LAM-003 300 mg QD | LAM-003 450 mg QD | LAM-003 600 mg QD
Number analyzed (Participants) | 6 | 3 | 4 | 4
ng/mL
  LAM-003A Day 1: number analyzed (Participants) | 5 | 3 | 1 | 4
  LAM-003A Day 1 | 3550 (1860) | 8360 (2230) | 9170 | 8240 (3750)
  LAM-003A Day 8: number analyzed (Participants) | 5 | 3 | 1 | 4
  LAM-003A Day 8 | 5000 (576) | 8360 (1150) | 8500 | 9620 (3810)
  LAM-003 Day 1: number analyzed (Participants) | 3 | 3 | 1 | 4
  LAM-003 Day 1 | 0.560 (0.320) | 1.47 (1.28) | 2.71 | 1.83 (1.30)
  LAM-003 Day 8: number analyzed (Participants) | 4 | 3 | 1 | 4
  LAM-003 Day 8 | 0.617 (0.220) | 1.08 (1.36) | 3.60 | 1.45 (1.43)

4. Secondary Outcome: Time of Maximum Concentration [Tmax]
Description: The pharmacokinetic parameter Tmax was determined in plasma for the active metabolite of LAM-003A and LAM-003 (prodrug)
Time Frame: Cycle 1 Days 1, 2 and 8 (1 cycle = 28 days)
Population: The PK population included all evaluable participants who were dosed and had sufficient concentration-time data to estimate at least one of the planned PK parameters, as determined by the study pharmacokineticist.
Measure: Median (Full Range); unit: hours
Arm/Group | LAM-003 200 mg QD | LAM-003 300 mg QD | LAM-003 450 mg QD | LAM-003 600 mg QD
Number analyzed (Participants) | 6 | 3 | 1 | 4
hours
  LAM-003A for Day 1: number analyzed (Participants) | 5 | 3 | 1 | 4
  LAM-003A for Day 1 | 3.80 [1.00 to 4.00] | 3.80 [1.80 to 4.00] | 4.10 [4.10 to 4.10] | 1.95 [1.90 to 23.3]
  LAM-003A for Day 8: number analyzed (Participants) | 5 | 3 | 1 | 4
  LAM-003A for Day 8 | 2.00 [1.80 to 4.00] | 4.00 [4.00 to 5.80] | 2.10 [2.10 to 2.10] | 1.95 [1.10 to 2.00]
  LAM-003 for Day 1: number analyzed (Participants) | 3 | 3 | 1 | 4
  LAM-003 for Day 1 | 1.00 [0.50 to 1.00] | 1.80 [0.80 to 2.00] | 0.50 [0.50 to 0.50] | 0.50 [0.40 to 1.00]
  LAM-003 for Day 8: number analyzed (Participants) | 4 | 3 | 1 | 4
  LAM-003 for Day 8 | 0.75 [0.50 to 1.00] | 1.10 [0.50 to 1.10] | 0.50 [0.50 to 0.50] | 1.10 [0.600 to 3.00]

5. Secondary Outcome: Area Under the Curve [AUC]
Description: The pharmacokinetic parameter area under the concentration-time curve was determined in plasma for the active metabolite of LAM-003A and LAM-003 (prodrug). AUClast is the area under the concentration-time curve from time-zero to the time of the last quantifiable concentration. AUCtau is the area under the concentration-time curve during the dosing interval where tau=24hours for once daily (QD) dosing. AUCtau was not calculated for LAM-003.
Time Frame: Cycle 1 Days 1, 2 and 8 (1 cycle = 28 days)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | LAM-003 200 mg QD | LAM-003 300 mg QD | LAM-003 450 mg QD | LAM-003 600 mg QD
Number analyzed (Participants) | 6 | 3 | 1 | 4
h*ng/mL
  LAM-003A AUClast for Day 1: number analyzed (Participants) | 5 | 3 | 1 | 4
  LAM-003A AUClast for Day 1 | 43100 (23200) | 112000 (45100) | 131000 | 105000 (39800)
  LAM-003A AUClast for Day 8: number analyzed (Participants) | 5 | 3 | 1 | 4
  LAM-003A AUClast for Day 8 | 24400 (5680) | 53600 (10400) | 52800 | 56400 (18000)
  LAM-003 AUClast for Day 1: number analyzed (Participants) | 3 | 3 | 1 | 4
  LAM-003 AUClast for Day 1 | 0.287 (0.254) | 0.958 (0.745) | 1.72 | 0.935 (1.10)
  LAM-003 AUClast for Day 8: number analyzed (Participants) | 4 | 3 | 1 | 4
  LAM-003 AUClast for Day 8 | 0.383 (0.311) | 1.18 (1.84) | 0.90 | 0.833 (0.837)
  LAM-003A AUCtau for Day 1: number analyzed (Participants) | 4 | 3 | 1 | 3
  LAM-003A AUCtau for Day 1 | 26000 (43900) | 113000 (46100) | 132000 | 110000 (47300)
  LAM-003A AUCtau for Day 8: number analyzed (Participants) | 3 | 0 | 1 | 4
  LAM-003A AUCtau for Day 8 | 42300 (4840) |  | 113000 | 103000 (33900)

6. Secondary Outcome: Objective Response Rate
Description: Tumor response by AML response criteria (Cheson 2003).
Time Frame: Every 8 to 12 weeks for up to 48 weeks.
Population: All participants who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LAM-003 200 mg QD | LAM-003 300 mg QD | LAM-003 450 mg QD | LAM-003 600 mg QD
Number analyzed (Participants) | 6 | 3 | 4 | 4
Participants
  CRc: Composite complete remission including participants with CR, CRMRD-, and CRi | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0
  Treatment Failure | 3 | 1 | 2 | 3
  Disease Relapse or Progression | 2 | 2 | 2 | 1
  Nonevaluable | 1 | 0 | 0 | 0

7. Secondary Outcome: Event-Free Survival (EFS) and Overall Survival (OS)
Description: Event-free survival (EFS), defined as the interval from the start of study therapy to the earliest of the first documentation of disease relapse, disease progression, treatment failure (TF), or death from any cause. Overall survival (OS), defined as the interval from the start of study therapy to death from any cause.
Time Frame: Every 8 to 12 weeks for up to 48 weeks.
Population: All participants who received ≥1 dose of study drug.
Measure: Median (Full Range); unit: months
Arm/Group | LAM-003 200 mg QD | LAM-003 300 mg QD | LAM-003 450 mg QD | LAM-003 600 mg QD
Number analyzed (Participants) | 6 | 3 | 4 | 4
months
  EFS | 0.6 [0.1 to 1.9] | 0.9 [0.7 to 1.2] | 1.8 [0.3 to 3.5] | 1.5 [0.6 to 2.9]
  OS | 3 [0.3 to 3.2] | 5.1 [1.0 to 5.9] | 3.4 [0.8 to 5.5] | 3.1 [1.6 to 4.3]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the signing of informed consent through to 30 days after the final dose of study drug administration or when any ongoing drug-related AEs and/or serious adverse events (SAEs) have resolved or become stable (up to Week 48).
Description: Adverse events are displayed by the dose group the participant was initially enrolled in, irrespective of intrasubject dose modifications.
Groups:
- LAM-003 450 mg QD: 4 participants were accrued at 450 mg QD.
- LAM-003 600 mg QD: 4 participants were accrued at 600 mg QD.
- LAM-003 750 mg QD: 3 participants received 750 mg QD after intrasubject dose escalations.
  • Subject 006-006 received LAM-003 450 mg QD during Cycles 1, 600 mg LAM-003 in Cycle 2 and received LAM-003 750 mg QD during Cycles 3 and 4.
  Subject 005-011 received LAM-003 600 mg QD during Cycle 1 and received LAM-003 750 mg QD during Cycles 2 and 3.
  • Subject 006-007 received LAM-003 600 mg QD during Cycle 1 and received LAM-003 750 mg QD during Cycle 2.
Arm/Group | LAM-003 200 mg QD | LAM-003 300 mg QD | LAM-003 450 mg QD | LAM-003 600 mg QD | LAM-003 750 mg QD
All-Cause Mortality (participants affected / at risk) | 2/6 | 1/3 | 2/4 | 1/4 | 2/3
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/3 | 3/4 | 2/4 | 2/3
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 4/4 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LAM-003 200 mg QD (N=6) | LAM-003 300 mg QD (N=3) | LAM-003 450 mg QD (N=4) | LAM-003 600 mg QD (N=4) | LAM-003 750 mg QD (N=3)
Disease Progression (General disorders) | 1 | 1 | 2 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0
Hemoglobin Decreased (Investigations) | 0 | 0 | 0 | 1 | 0
WBC Count Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Cerebral Hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hemorrhage Intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LAM-003 200 mg QD (N=6) | LAM-003 300 mg QD (N=3) | LAM-003 450 mg QD (N=4) | LAM-003 600 mg QD (N=4) | LAM-003 750 mg QD (N=3)
Oedma peripheral (General disorders) | 3 | 2 | 0 | 1 | 1
Pyrexia (General disorders) | 2 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 0 | 2 | 1
Chills (General disorders) | 1 | 2 | 1 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 1 | 0 | 0
Pain (General disorders) | 2 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 2 | 1 | 1 | 1 | 0
Platelet count decreased (Investigations) | 4 | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 4 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 1 | 0 | 1 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 1 | 0
Hemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Tropoin T increased (Investigations) | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Plural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Decreased appetitie (Metabolism and nutrition disorders) | 2 | 2 | 2 | 2 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 2 | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Pallor (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Anal abcess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hypobarism (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eyelid pain (Eye disorders) | 0 | 1 | 0 | 0 | 0
Leukaemia cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Scrotal irritation (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT03426605/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT03426605/SAP_001.pdf